CLINICAL TRIAL: NCT07144657
Title: Prospective Study of Frontline Antibiotics Therapy in the Treatment of Early-stage Helicobacter Pylori-negative Gastric Mucosa-associated Lymphoid Tissue Lymphoma
Brief Title: Prospective Study of Frontline Antibiotics Therapy in the Treatment of Early-stage HP-negative Gastric MALT Lymphoma
Acronym: GastricMALToma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, Professor and Attending Physician, National Taiwan University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202410042MINE; NTUH (Other: Department of Oncology, National Taiwan University Hospital)
Record Dates: First submitted 2025-06-18; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-06

CONDITIONS: MALT Lymphoma of Stomach
Keywords: Helicobacter pylori-negative; MALT lymphoma; Stomach; Clarithromycin; Antibiotics treatment; Low-dose cyclophosphamide
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone | interventions — Esomeprazole; bismuth tripotassium dicitrate; Tetracycline; Metronidazole; Clarithromycin; Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: 1. Frontline antibiotics treatment (two weeks of quadruple HPE regimens followed by 4 weeks of oral clarithromycin) The 14 days regimen of quadruple HPE regimens [40] Nexium (esomeprazole) 40 mg 1# bid PO Days 1-14 Bismuth tripotassium dicitrate 300 mg 1# qid PO Days 1-14 Tetracycline 500 mg 1# qid PO Days 1-14 Metronidazole 500 mg 1# tid PO Days 1-14 4 weeks of single agent clarithromycin following quadruple HPE regimens Clarithromycin 500 mg 1# bid PO Days 15-42
  2. Second line immune-modulator regimens (CAMC, clarithromycin (CAM) and low-dose cyclophosphamide) for antibiotics-unresponsive HP-negative gastric MALT lymphoma 2.1 Oral clarithromycin (CAM) once daily for 21 days at a dose 500 mg. 2.2 Oral cyclophosphamide (Endoxan) once daily for 21 days at a dose 50 mg.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The treatment efficacy of antibiotics treatment (Experimental): 1. Frontline antibiotics treatment (two weeks of quadruple HPE regimens followed by 4 weeks of clarithromycin).
  2. Second line immune-modulator regimens (CAMC, clarithromycin (CAM) and low-dose cyclophosphamide) for antibiotics-unresponsive HP-negative gastric MALT lymphoma.
  Interventions: Drug: Esomeprazole, Bismuth tripotassium dicitrate, Tetracycline, and Metronidazole

INTERVENTIONS:
Drug: Esomeprazole, Bismuth tripotassium dicitrate, Tetracycline, and Metronidazole — 1. Frontline antibiotics treatment (two weeks of quadruple HPE regimens followed by 4 weeks of clarithromycin).
  2. If no response to frontline antibiotics treatment, second line immune-modulator regimens (CAMC, clarithromycin (CAM) and low-dose cyclophosphamide) will be prescribed
  Other Names: Clarithromycin; Cyclophosphamide

SUMMARY:
We hypothesized that a proportion of patients with localized Helicobacter pylori-negative gastric MALT lymphoma may well respond to frontline Helicobacter pylori eradication therapy (HPE) and remain lymphoma-free for the long term. In addition, we hypothesized that for patients with antibiotics-unresponsive HP-negative gastric MALT lymphoma, the administration of a combination of clarithromycin and low-dose cyclophosphamide (CAMC) could result in tumor regression through the direct anti-neoplastic effects and the indirect immune modulatory effect.

Therefore, in this proposal, we will design a prospective phase II study to evaluate the treatment efficacy of frontline HPE, consisting of two weeks of quadruple HPE regimen followed by four weeks of clarithromycin in patients with stage IE/IIE1 HP-negative gastric MALT lymphoma. In addition, we will treat patients who did not respond to HPE using combination regimens of clarithromycin and low-dose cyclophosphamide (CAMC).

DETAILED DESCRIPTION:
Gastric mucosa-associated lymphoid tissue (MALT) lymphoma (marginal zone B-cell lymphoma) is the most common extranodal MALT lymphoma. Since the association between Helicobacter pylori (HP) infection and gastric and duodenal ulcers, the administration of antibiotics plus proton pump inhibitors (PPIs) eradicating HP has been reported to cure the disease of ulcers and decrease the incidence of subsequent gastric cancer. The prevalence of HP-positive gastric MALT lymphoma has decreased over the last two decades, whereas that of HP-negative gastric MALT lymphoma has increased. For example, Raderer et al. showed an increased prevalence of HP-negative infection in patients with gastric MALT lymphoma diagnosed after 2004 compared with those diagnosed before 2004 (31.2% versus 18%; a total of 97 cases). Mendes et al. also found that the prevalence of HP-negative infection in gastric MALT lymphoma diagnosed between 2005 and 2013 was 67.6% (25/37).

In contrast to most HP-positive gastric MALT lymphomas that respond to frontline HP eradication therapy (HPE), the efficacy of frontline antibiotics in the treatment of HP-negative gastric MALT lymphomas remains ambiguous. Several case series reported that a proportion of patients with localized HP-negative gastric MALT lymphoma can be cured by a frontline HPE-like regimen. Between January 1, 2005, and June 30, 2014, we reviewed 25 patients with newly diagnosed stage IE/IIE1 primary HP-negative gastric MALT lymphoma who underwent frontline HPE-like regimen, which consist of 500 mg of amoxicillin administered four times a day (or 1000 mg of amoxicillin administered twice a day), 500 mg of clarithromycin administered twice a day, and 20 mg of omeprazole or 30 mg lansoprazole administered twice a day for 2 weeks as frontline treatment. An HP-negative status was defined as total negative results on histology (including HP, atrophic gastritis, and intestinal metaplasia), a rapid urease test, a 13C urea breath test, and serology. Based on the criteria of Groupe d'Etude des Lymphomes de l'Adult (GELA) for tumor response, we observed antibiotic responses in 9 (36.0%; 95% confidence interval [CI], 17.2-54.8%; complete remission [CR], n = 8; partial remission [PR], n = 1) out of 25 patients, and the median time to a CR was 7 months (95% CI, 0.1-13.9 months). Of 20 patients receiving serum immunofixation electrophoresis (IFE) assessments, immunoglobulin M lambda monoclonal gammopathy was detected in 3 (25.0%) of the 12 antibiotic-unresponsive tumors, but not in the 8 antibiotic-responsive tumors (p = 0.242). At a median follow-up of 51.0 months (95% CI, 34.7-67.3 months), all patients with responsive tumors after HPE therapy were alive and free of lymphomas and progression.

In addition to eradicating HP and HP-like bacteria, clarithromycin has been reported to have an effect in the cure of a proportion of extragastric MALT lymphoma. Ferreri et al. reported that high-dose clarithromycin (2 g a day for 14 days for each course) resulted in a CR rate of 26.9% in patients with relapsed or refractory extranodal MALT lymphoma. In a B-cell lymphoma cell line derived from a BALB/c mouse model, O'Hara et al. showed that clarithromycin inhibited cell viability and induced apoptosis through down-regulating Bcl-2 expression. Mizunoe et al. showed that macrolides, either clarithromycin (100 ug/ml) or azithromycin (100 ug/ml), caused apoptosis of activated lymphocytes via Annexin-V analyses, and the effect of augmentation of apoptosis is through attenuation of Bcl-xL expression. Another macrolide, erythromycin, was found to have an inhibitory effect on the proliferation of human Jurkat T cells, and a possible mechanism is the down-regulation of NF-kB expression. In CD4+ T-cells, azithromycin effectively inhibited cell proliferation and cytokine secretion through down-regulation of the activity of mammalian target of rapamycin (mTOR). The aforementioned immunosuppressive effect on CD4+ T-cells was also observed at a higher concentration of clarithromycin (40 mg/L). At 40 mg/L of azithromycin and clarithromycin, secretion of cytokines, such as IL-2, IL-10, IL-13, IL-17, and IFN-gamma, was reduced in their study.

For patients with antibiotic-unresponsive MALT lymphoma, several new drugs, including bendamustine, bortezomib, and new compounds of alkylating agents, have been demonstrated to provide approximately 50% ORR but result in grade III/IV myelosuppression. Therefore, it is important to seek biological agents that provide excellent efficacy and result in fewer adverse effects for these patients (since most patients are older). Considering that most patients with MALT lymphoma are newly diagnosed at an older age, our pilot study evaluates the efficacy of low-dose single chlorambucil or low-dose single cyclophosphamide in patients with antibiotic-unresponsive MALT lymphoma. We reported that a single low-dose cyclophosphamide (50 mg daily for 21 days, every 28 days) alone resulted in the ORR of 44.4 % in 9 patients with antibiotic-unresponsive MALT lymphoma. In addition to killing lymphoma cells, single low-dose cyclophosphamide (i.e., 25-100 mg in adults), is an option for restoring immune response in patients with advanced cancer. The main mechanism of cyclophosphamide in counteracting immunosuppression in cancer is the result of selective suppression of regulatory T cells (Tregs) and restoration of T and natural killer (NK) effector functions.

Considering that clarithromycin and low-dose cyclophosphamide are found to have anti-tumor effects and immune-modulatory effects in MALT lymphoma in our and other investigators' results, we speculated that combined clarithromycin and low-dose cyclophosphamide can increase the ORR rate as well as durable tumor remission and decrease aggressive chemotherapy-related adverse effects in antibiotic-unresponsive HP-negative gastric MALT lymphoma. Therefore, in this proposal, we will design a prospective phase II study to evaluate the treatment efficacy of frontline bismuth-based quadruple therapy of HPE regimens followed by 4 weeks of clarithromycin in patients with HP-negative gastric MALT lymphoma. In addition, we investigate whether the combined clarithromycin and low-dose cyclophosphamide (combined regimen: CAMC) is an effective regimen for targeting patients with antibiotic-unresponsive HP-negative gastric MALT lymphoma. We will explore the potential biological markers to predict the antibiotic's responsiveness and the responses of CAMC in this project.

We hypothesized that a proportion of patients with localized HP-negative gastric MALT lymphoma may well respond to frontline HPE and remain lymphoma-free for the long term. In addition, we hypothesized that for patients with antibiotics-unresponsive HP-negative gastric MALT lymphoma, the administration of a combination of clarithromycin and low-dose cyclophosphamide (CAMC) could result in tumor regression through the direct anti-neoplastic effects and the indirect immune modulatory effect.

Therefore, in this proposal, we will design a prospective phase II study to evaluate the treatment efficacy of frontline HPE, consisting of two weeks of quadruple HPE regimen, including esomeprazole 40 mg 1# bid PO Days 1-14, bismuth tripotassium dicitrate 300 mg 1# qid PO Days 1-14, tetracycline 500 mg 1# qid PO Days 1-14, and metronidazole 500 mg 1# tid PO Days 1-14, followed by four weeks of clarithromycin in patients with stage IE/IIE1 HP-negative gastric MALT lymphoma. In addition, we will treat patients who did not respond to HPE using combination regimens of CAMC.

ELIGIBILITY:
Inclusion Criteria:

1. The patients must have histologically confirmed primary gastric MALT lymphoma by REAL/WHO classification
2. The patient must have no prior chemotherapy or radiotherapy for his/her gastric MALT lymphoma
3. Patients must have evaluable disease by endoscopy and/or the nodal status by computed tomography 3.1 If patients have endoscopic lesions without computed tomography-demonstrating lesions are eligible.

   3.2 Endoscopic ultrasonography (EUS) is optional to evaluate the depth of tumor infiltration and for status of perigastric lymph node enlargement
4. Patients must have documented to have no HP infection before treatment, which will be evaluated by the following tests: histology, rapid urease test (CLO-test), C-13 urease breath test, HP stool antigen, and serology; and all of the five tests have to be negative for the diagnosis of no evidence of HP infection.
5. Patients must have either stage IE or IIE1 disease, according to an adaptation of the Ann Arbor staging system modified by Musshoff for primary extranodal lymphoma.
6. Patients must have signed the informed consent and agree to provide achieved pathologic material and tumor biopsy for translational study
7. Patients must have signed the informed consent and agree to provide achieved blood samples for potential serum molecular studies and fecal samples for researches of gut microbiota

Exclusion Criteria:

1. Active second malignancies during the last five years except non melanomatous skin cancer, carcinoma in situ of cervix, lobular or ductal carcinoma in situ of breast.
2. Patients with previous history of extranodal lymphoma are not eligible.
3. Patients with stage IIE2 or beyond disease: infiltration of regional lymph nodes not adjacent primary involved site.
4. Patients with cardiopulmonary status that do not allow repeat examination are not eligible.
5. Patients with prior chemo- or radiotherapy for their extragastric lymphoma are not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
The treatment efficacies of frontline antibiotics treatment for Helicobacter pylori-negative gastric MALT lymphoma | 2 years
  1. The overall response rate (including complete remission [CR] and partial remission [PR]) for frontline antibiotics treatment (two weeks of quadruple HPE regimens followed by 4 weeks of clarithromycin) in stage IE/IIE1 HP-negative gastric MALT lymphoma.
  2 The median time to CR or PR after completion of antibiotics and duration of CR or PR.
  3 The overall response rate (including CR and PR) for immune treatment (CAMC) in antibiotics-unresponsive HP-negative gastric MALT lymphoma

SECONDARY OUTCOMES:
The clinical outcomes of HP-negative gastric MALT lymphoma after antibiotics treatment and low-dose cyclophosphamide and clarithromycin | 3 years
  1. The event-free survival and overall survival of all patients.
  2. The biological markers in predicting the antibiotic-responsiveness of HP- negative gastric MALT lymphoma
  3. The biological markers in predicting the CAMC-responsive of antibiotics- unresponsive HP-negative gastric MALT lymphoma
  4. The assessment of adverse effects of CAMC immune regimen.
  5. The identification of microbiota, including non-Helicobacter pylori Helicobacter (NHPH), the other bacteria, or gut microbiota that contributes to the lymphomagenesis of HP-negative gastric MALT lymphoma

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, None Selected, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
Wait for the actual enrollment and the completion of this phase II trial